CLINICAL TRIAL: NCT02468869
Title: Improving Discharge Communication in the Emergency Department Through Information Structuring: A Cluster Randomized Controlled Trial
Brief Title: Improving Discharge Communication in the Emergency Department Through Information Structuring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: University of Basel (Other); Max Planck Institute for Human Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: BACOP2
Record Dates: First submitted 2015-05-27; First posted 2015-06-11 (Estimated); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Information Structuring Skills; Empathy Skills
Keywords: Recall; Discharge communication; Satisfaction; Adherence; Information structuring; Empathy skills
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Information structuring skills training (Experimental): Physicians received a communication skills training focusing on information structuring with the so-called book metaphor for a structured discharge communication with the patient.
  Interventions: Behavioral: Communication skills training "information structuring skills"
- Empathy skills training (Active Comparator): Physicians received a communication skills training focusing on empathy skills with the acronym NURSE for an empathetic discharge communication with the patient.
  Interventions: Behavioral: Communication skills training "empathy skills"

INTERVENTIONS:
Behavioral: Communication skills training "empathy skills"
  Arms: Empathy skills training
Behavioral: Communication skills training "information structuring skills"
  Arms: Information structuring skills training

SUMMARY:
The goal of the proposed study is to assess the potential of information structuring for improving discharge communication. Specifically, the investigators aim to examine the advantages of an information-structuring skills training for physicians (compared to an empathy skills training) on discharge communication and associated patient outcomes, such as patients' information recall and adherence to physician recommendations. The investigators hypothesize that patients receiving structured discharge information from their trained physicians will be able to recall more information and show higher adherence to recommendations relative to controls (i.e., patients receiving discharge information from doctors trained in empathy skills).

ELIGIBILITY:
Inclusion Criteria:

* Outpatients with chest pain
* Outpatients with abdominal pain

Exclusion criteria:

* Patients younger than 18 years of age (limited ability to provide informed consent)
* Patients with limited ability to communicate in German, the default language at the hospital (confounder related to language proficiency)
* Patients with dementia (confounder arising from pathological memory deficits)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Patients' recall of the information provided during discharge communication | 3 times: immediately after discharge, one week after discharge, one month after discharge

SECONDARY OUTCOMES:
Adherence to recommendations | 2 times: one week and one month after discharge
Patient satisfaction in four dimensions | Immediately after discharge
  (1) comprehension, (2) structuredness (3) recommendation of the physician to family and friends (4) informativeness

CONTACTS AND LOCATIONS:
Overall Officials: Roland Bingisser, Prof. Dr., Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Emergency Department, Basel, Canton of Basel-City, Switzerland